CLINICAL TRIAL: NCT01972997
Title: A Single-center, Randomized, Double-blinded, Prospective Study to Assess the Changes in the 24-hour IOP (Intraocular Pressure) Pattern in Relation to SENSIMED Triggerfish® Sensor Sizes in Healthy Subjects
Brief Title: SENSIMED Triggerfish Sensor Sizes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: TF-1220
Record Dates: First submitted 2013-07-26; First posted 2013-10-31 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- SENSIMED Triggerfish (Experimental): There is only 1 arm in the study. SENSIMED Trigerfish lens sensors with different base curves are placed on subjects in random and double-blinded manner in sequential sessions.
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish

SUMMARY:
This is a study investigating the effect of various SENSIMED Triggerfish sensor lens sizes on the recorded IOP related patterns in 10 healthy volunteers. Each volunteers receives 4 24-hours sessions of pattern recording on one selected eye (study eye). Each of the sensor lens sizes is placed on the eye in the different sessions. Subjects visit the study site for installation and removal of the device and accompanying exams, but remain ambulatory during the recording.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject without previous ocular disease
* Aged ≥ 18 years, of either sex
* Central corneal radius (flat meridian) between 7.75 mm and 8.25 mm in at least one eye
* Not more than 6 diopters spherical equivalent in the study eye
* Having given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Subjects with allergy to corneal anesthetic
* Subjects with contraindications for silicone contact lens wear
* Subjects not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Any other contra-indication listed in the TF user manual

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The effect of the sensor lens size on IOP patterns as recorded by TF (SENSIMED Triggerfish) as compared to the recommended sensor lens fit | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain